CLINICAL TRIAL: NCT04061187
Title: Livestreaming From Smartphones as a Supplement to Emergency Calls
Status: Completed | Type: Observational
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: The Danish foundation TrygFonden (Unknown)
Responsible Party: Sponsor
Other Study IDs: F-35150-03
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Emergencies; Unconscious
Keywords: Dispatcher; Dispatcher-assisted cardiopulmonary resuscitation; Emergency call; Live video
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Emergencies; Unconsciousness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to analyse if live video as a supplement to emergency calls can improve medical dispatchers' situation awareness and enhance the assistance they provide including provision of pre-hospital resources. Focus will also be on evaluating the unconscious patient and improve CPR quality.

The general experience from the medical dispatcher and the person calling the emergency number regarding the feasibility of adding live video will also be analysed.

DETAILED DESCRIPTION:
Setting; The study will be conducted in Copenhagen Emergency Medical Services (EMS), which covers a population of approximately 1.84 million people and an area of 2559 km2. In case of an emergency, there is a single emergency phone number (1-1-2) to a call center that identifies the need for police, fire or medical assistance. If the problem is medical, the caller is re-directed to the EMS where medical dispatchers answer, process and respond to the call by activating the appropriate EMS response and delivering medical advice.

In every emergency call, the medical dispatcher starts by asking the caller about the nature of the problem and whether the patient is awake and breathing normally. In case of suspected cardiac arrest, the dispatcher follows a guideline for dispatcher assisted cardiopulmonary resuscitation based on the European Resuscitation Council Guidelines for Resuscitation. The medical dispatchers are specially trained registered nurses or paramedics with experience within emergency care. They all have a basic life support course and advanced course in DA-CPR. Their decision-making process is supported by a criteria-based, nationwide Emergency Medical Dispatch System (Danish Index), which is a validated tool for managing emergency calls for the most urgent cases of emergencies. The instructions in DA-CPR is divided into two depending on whether the bystander have received a basic CPR course (BLS course). If the bystanders have a BLS course they are also instructed in ventilation. Instructions to lay people consist of short commands. E.g., "place the victim in the supine position". All medical dispatcher has a metronome available to support they guidance. The medical dispatcher guide bystander until ambulance arrival.

Methods; When the medical dispatcher receives an emergency call they decide emergency priority level, dispatch vehicle type and competence allocation and guide in CPR as before the study. Afterwards then can add livestreaming to the emergency call. Each medical dispatcher can choose in which emergency call they want to add live video, but they are recommended to do it with all unconscious patients including cardiac arrest after bystander CPR is started.

Technical solution; For livestreaming of video footage the dispatcher sends a text message, asking the caller to give their consent to share stream video from their camera on their smartphone. When the caller confirms consent, the smartphone automatically starts securely transmitting a video live stream from the scene back to the medical dispatcher. When the emergency call is finished the link will be inactivated.

Data collection and outcome; All medical dispatchers will participate. After each emergency call with stream of live video the medical dispatcher fills out a questionnaire about their evaluations of the patient before and after live video, if the live video resulted in changed treatment of the patient, or different response. Emergency priority level, emergency response, date and time for the call and symptom-based criteria from Danish Index (1-39 items) will be collected from the dispatch system Logis CAD and compared with emergency calls without use of live video.

The person calling the emergency number 1-1-2 and accepted transmission of live video to the emergency medical dispatcher will afterwards receive a text message with a questionnaire about their experience. We will collect data for aprox. 500 emergency calls where live video is added to the call including around 200 cases with unconscious patients and 53 cases with cardiac arrest patients. We will analyse the change in CPR quality before the medical dispatcher assist in CPR using live video and after the medical dispatcher has assisted. The first evaluation of CPR quality will be as soon as possible from the streamed video and the after score will be registered when the CPR is optimized as much as possible.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion criteria (stream live video footage) These are assessed by the medical dispatcher before stream of live video footage.

* Emergency call about an unconscious patient. (The patient is defined as unconscious, if the patient is unresponsive to verbal or pain stimulus according to the Danish Index. (Inclusion criterion in relation to the Danish Index is "unconscious patient with normal breathing. A.01.03", as well as all sub-criteria that meet the above criteria e.g. "A.06.01, Unresolved problem;" Does not respond to call or pain stimulus, but no breathing problems ").
* Emergency call about suspected cardiac arrest where CPR is provided
* Emergency call about a patient with trauma/illness where the medical dispatcher thinks it will be a benefit with live video footage
* Video-capable smartphone present
* Caller by the patient's side
* Caller expected age≥ 18 years
* More than two bystanders present

Exclusion Criteria:

* If caller, patient or other bystanders do not want livestreaming to be added to the emergency call.
* No video-capable smartphone present
* Caller not by the patient's side
* Caller a child
* Less than two bystanders present

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Emergency medical dispatchers in Copenhagen who added live video footage to the emergency call
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Changed emergency response after adding live video to the emergency call | From the beginning of the emergency call to the end of the call. Approx. 6-7 minutes
  Did the medical dispatcher change emergency response more often after live video was added to the emergency call compared to emergency calls without video.
The medical dispatcher's evaluations of the patient after adding live video footage to the emergency call. | From the beginning of the emergency call to the end of the call. Approx. 6-7 minutes
  Did the medical dispatcher's evaluation of the patient change because of the live video footage? (ANSWER: Yes, patient more critical ill/ Yes, less critical ill/ or no change) Did the patient suffer another trauma/disease compared to what the medical dispatcher thought before the live video footage? (ANSWER: No/Yes (describe)).
The medical dispatcher's evaluations of the patient's level of consciousness before and after adding live video footage to the emergency call. | From the beginning of the emergency call to the end of the call. Approx. 6-7 minutes.
  The medical dispatcher evaluate the patient's level of consciousness before and after the live video footage; AVPU scale (an acronym from "alert, verbal, pain, unresponsive") /or inaccessible.
The medical dispatcher's evaluations of the surroundings and bystander response after adding live video footage to the emergency call. | From the beginning of the emergency call to the end of the call. Approx. 6-7 minutes.
  Did the medical dispatcher situation's awareness regarding the surroundings or bystander response change after video footage? (ANSWER: No/ Yes, Less bystanders present/ Yes, more bystanders present/ Yes, bystander response were more sufficient/ Yes, bystander response were less sufficient/Yes, surroundings were different(describe)/ other (describe)).
The medical dispatcher's evaluations of the usefulness of adding live video footage to the emergency call. | From the beginning of the emergency call to the end of the call. Approx. 6-7 minutes.
  Was the live video footage useful for the medical dispatcher"? (ANSWER: Extremely useful/ very useful/ moderately useful/ slightly useful/ not at all useful).
Change in emergency level after adding live video footage to the emergency call. | Evaluated at the end of the emergency call.
  Did the medical dispatcher change emergency priority level because of the live video footage?" (ANSWER: No, Yes (upgrade, downgrade))
Change in the CPR quality (hand position) before the medical dispatcher assist in CPR using the video footage (video-DA-CPR) and after the medical dispatcher has assisted . | From the medical dispatcher receive video footage until the end of video-DA-CPR.
  Correct hand position before and after video-DA-CPR? (Outcome: yes / no / inaccessible evaluated before and after video-DA-CPR)
Change in the CPR quality (compressions rate) before and after video-DA-CPR. | From the medical dispatcher receive video footage until the end of video-DA-CPR.
  Correct compressions rate (100-120 compressions/min) before and after video-DA-CPR (Outcome: yes / no / inaccessible evaluated before and after video-DA-CPR)
Change in the CPR quality (compressions depth) before and after video-DA-CPR | From the medical dispatcher receive video footage until the end of video-DA-CPR.
  Correct compressions depth before and after video-DA-CPR (approximately one third of the anterior-posterior diameter). (Outcome: yes / no / inaccessible evaluated before and after video-DA-CPR)

SECONDARY OUTCOMES:
"Hands-of-time" during CPR | From the medical dispatcher receive video footage until the end of the call. Approx. 5-6 minutes.
  Does the medical dispatcher initiate less "hands-of-time" during CPR after receiving live video footage? "Hands-off-time" is the time with no chest compressions. (ANSWER: does the dispatcher initiate less "hands-of-time"?(yes/No))
Ventilations performed by bystanders? | From the medical dispatcher receive video footage until the end of video-DA-CPR.
  Correct ventilations before and after video-DA-CPR? (Outcome: yes / no / inaccessible evaluated before and after video-DA-CPR).
Shift of persons during CPR | From the medical dispatcher receive video footage until the end of the call. Approx. 5-6 minutes.
  Shift of persons during CPR? (Outcome:yes/no), does bystander initiate this by themselves or guide by the dispatcher?
Use of AED | From the medical dispatcher receive video footage until the end of the call. Approx. 5-6 minutes.
  Correct attachment of AED pads (Outcome:yes/no), If "no" does the dispatcher initiate correct use?
Other aspects of bystander CPR | From the medical dispatcher receive video footage until the end of the call. Approx. 5-6 minutes.
  Did the dispatcher assist in other aspects of CPR? (describe)
Bystanders experiance with adding live video to the emergency call | From the person calling 1-1-2 accept transmission of live video until end of the call. Approx. 5-6 minutes.
  Bystanders' evaluation of the potential help and challenges with adding live video to the emergency call

CONTACTS AND LOCATIONS:
Overall Officials: Freddy K. Lippert, MD, CEO, Principal Investigator — Copenhagen Emergency Medical Services; Fredrik Folke, MD, PhD, Study Chair — Copenhagen Emergency Medical Services; Christian S. Meyhoff, MD, PhD, Study Chair — Department of Anaesthesia and Intensive Care, Bispebjerg and Frederiksberg Hospital, Denmark; Doris Øestergaard, MD, Prof., Study Chair — Copenhagen Academy for Medical Education and Simulation, Denmark.; Gitte Linderoth, MD, Study Director — Copenhagen Emergency Medical Services
Locations (1):
- Copenhagen Emergency Medical Services, Copenhagen, Ballerup, Denmark

IPD SHARING:
Plan to Share IPD: No